CLINICAL TRIAL: NCT00826956
Title: The Changes of Pulmonary Blood Flow in Nondependent Lung During One Lung Ventilation
Brief Title: The Change of Pulmonary Blood Flow During One Lung Ventilation
Status: Temporarily not available | Type: Expanded Access
Sponsor: Sichuan University (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Wei Wei, Department of Anesthesiology, West China Hospital, Sichuan University.
Other Study IDs: 30672026
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: One Lung Ventilation
MeSH Terms: interventions — One-Lung Ventilation

INTERVENTIONS:
Procedure: one lung ventilation — measure the pulmonary blood flow in nondependent lung during 30min one lung ventilation

SUMMARY:
To investigate the changes of regional pulmonary blood flow in nondependent lung by transesophageal echocardiography during one lung ventilation

ELIGIBILITY:
Inclusion Criteria:

* adult patients (ASA physical status I-III) requiring OLV for selective thoracic surgery.

Exclusion Criteria:

* chronic obstructive pulmonary disease
* hypertension
* cardiovascular
* esophageal disease

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Wang M, Gong Q, Wei W. Estimation of shunt fraction by transesophageal echocardiography during one-lung ventilation. J Clin Monit Comput. 2015 Apr;29(2):307-11. doi: 10.1007/s10877-014-9606-2. PMID 25155453